CLINICAL TRIAL: NCT01987141
Title: WATE Study - Gestational Weight Gain and the Electronic Medical Record
Brief Title: Gestational Weight Gain and the Electronic Medical Record
Acronym: WATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Scott Graziano, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205512
Record Dates: First submitted 2013-10-29; First posted 2013-11-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMR intervention (Experimental): Patients will have an electronic medical record popup/highlight in their chart, displaying the recommended guidelines for weight gain in pregnancy.
  Interventions: Other: EMR Intervention
- Control (No Intervention): The patient's medical record will be displayed as usual, with no flag or highlight for weight gain recommendations

INTERVENTIONS:
Other: EMR Intervention — Electronic medical record flag/notification in the patient's chart
  Arms: EMR intervention

SUMMARY:
Less than one third of pregnant women actually achieve the Institute of Medicine's (IOM) recommended weight gain. To date, there are no randomized controlled trials studying the use of the electronic medical record to alert providers to initiate the counseling of patients on the IOM gestational weight gain recommendations.

In the investigator's planned study intervention, using the EPIC EMR system, an electronic alert (Best Practice Advisory) will appear for providers at each prenatal care visit. This alert will remind providers to counsel patients on the recommendations for gestational weight gain. The control group will receive standard prenatal care, without electronic alerts generated regarding BMI and gestational weight gain.

The investigators hypothesize that a higher percentage of patients who receive the intervention will meet the IOM guidelines for weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with a single intrauterine gestation
* Present for new OB visit up to 13 weeks and 6 days gestation

Exclusion Criteria:

* They have a multiple gestation pregnancy
* They are under the age of 18
* They do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight gain | At delivery, average of 40 weeks from enrollment
  Primary outcome will be measured as the percent of patients who achieve their recommended weight gain goal in pregnancy (IOM guidelines)

SECONDARY OUTCOMES:
Patient perception | At end of pregnancy, average of 40 weeks from enrollment
  Survey to patients at the end of pregnancy regarding how patients perceive and are influenced by EMR notifications and counseling

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States